CLINICAL TRIAL: NCT04854694
Title: Product Testing of the FaceView Mask™: Usability Survey
Status: Completed | Type: Observational
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Other Study IDs: 262478
Record Dates: First submitted 2021-04-16; First posted 2021-04-22 (Actual); Results first posted 2025-04-10 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-03

CONDITIONS: Hearing Disability
Keywords: lip reading; face mask

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- All Subjects: All participants will be fit tested for the masks to ensure that the appropriate size is used. Some participants will wear the FaceView Mask™ (first) for 5 minutes before wearing the conventional surgical N95 respirator for 5 minutes. Others will wear the conventional surgical N95 respirator (first) for 5 minutes before wearing the FaceView Mask™ for 5 minutes.
  All subjects will complete the study survey after exposure to the interventions.
  Interventions: Device: FaceView Mask™; Device: conventional surgical N95 respirator

INTERVENTIONS:
Device: FaceView Mask™ — transparent surgical N95 respirator designed to improve communication
Device: conventional surgical N95 respirator — standard N95 respirator

SUMMARY:
The study aims to gather participants' perceptions of the novel transparent surgical N95 respirator vs. a conventional surgical N95 respirator. Following fitting of the masks, participants will complete a questionnaire to provide their perceptions of fit, comfort, ease of use, and benefit to communication.

DETAILED DESCRIPTION:
The investigators will recruit adult participants to complete a usability survey on a transparent surgical N95 respirator (i.e., FaceView mask) designed to improve communication. The study aims to gather participants' perceptions of the novel transparent surgical N95 respirator vs. a conventional surgical N95 respirator. Following fitting of the masks (5 minutes wear time each), the participants will complete a questionnaire to provide their perceptions of fit, comfort, ease of use, and benefit to communication.

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years old
* have no health conditions that would prevent them from safely wearing an N95 respirator (e.g., severe asthma, chronic obstructive pulmonary disease)
* read in English and communicate in English or American Sign Language
* be able to provide or arrange their own transportation to the study location

Exclusion Criteria:

* Children are to be excluded from the proposed research project because the current FaceView Mask™ is designed for adults
* Adults who are non-English communicators
* Any adult with health conditions that would prevent them from safely wearing an N95 respirator (e.g., severe asthma, chronic obstructive pulmonary disease)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A goal of 200 participants is desired with a minimum of 125 to meet study targets. We will be contacting known persons (not cold contacts) with ability to share study brochure by e-mail:
  1. across the UAMS campus (e.g., College Deans, Center Directors, Program Directors);
  2. surrounding clinics;
  3. American Sign Language interpreter education at the University of Arkansas at Little Rock (Program Director)
  4. Arkansas School for the Deaf (Superintendent and/or Assistant to the Superintendent); and
  5. Communications Plus+ Interpreter Services, Inc. (owner and operator)
Sampling Method: Probability Sample
Enrollment: 202 (Actual)
Dates: Start 2022-11-15 (Actual); Primary Completion 2024-02-29 (Actual); Study Completion 2024-02-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Samuel R Atcherson, PhD, Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Transparent Mask First, Then Non-Transparent Mask: Participants completed fit testing protocol using the transparent mask first, followed by the same fit testing protocol with a non-transparent mask, then completed a questionnaire.
- Non-Transparent Mask First, Then Transparent Mask: Participants completed fit testing protocol using the non-transparent mask first, followed by the same fit testing protocol with a transparent mask, then completed a questionnaire.
Period: Overall Study
Arm/Group | Transparent Mask First, Then Non-Transparent Mask | Non-Transparent Mask First, Then Transparent Mask
Started | 101 | 101
Completed | 101 | 101
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Subjects: All participants will be fit tested for the masks to ensure that the appropriate size is used. Some participants will wear the FaceView Mask™ (first) for 5 minutes before wearing the conventional surgical N95 respirator for 5 minutes. Others will wear the conventional surgical N95 respirator (first) for 5 minutes before wearing the FaceView Mask™ for 5 minutes.
  All subjects will complete the study survey after exposure to the interventions.
  FaceView Mask™: transparent surgical N95 respirator designed to improve communication
  conventional surgical N95 respirator: standard N95 respirator
Arm/Group | All Subjects
Number analyzed (Participants) | 202
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 198
  >=65 years | 4
Age, Continuous [Mean (Full Range); unit: years] | 34.3 [18 to 72]
Sex/Gender, Customized [Count of Participants; unit: Participants] — Female, Male, Intersex, Prefer Not to Say
  Participants
    Female | 173
    Male | 28
    Intersex | 1
    Prefer Not to Say | 0
Sex: Female, Male [Count of Participants; unit: Participants] — At the outset of the study, we permitted participants to select male, female, intersex, or prefer not to say. Population: One participant identified as Intersex
  Participants
    number analyzed (Participants) | 201
    Female | 173
    Male | 28
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Ease of Understanding Another Person
Description: As recorded on the survey
  1. Difficult
  2. Somewhat difficult
  3. Somewhat easy
  4. Easy
Time Frame: 1 day
Measure: Count of Participants; unit: Participants
Groups:
- Transparent Mask: Wore FaceView Mask which is the transparent mask
- Non-Transparent Mask: Wore 3M N95 mask which is the non-transparent mask
Arm/Group | Transparent Mask | Non-Transparent Mask
Number analyzed (Participants) | 202 | 202
Participants
  Difficult | 0 | 24
  Somewhat difficult | 4 | 67
  Somewhat easy | 36 | 47
  Easy | 162 | 64

2. Secondary Outcome: Fit of the Mask
Description: As recorded on the survey
  1. Extremely small
  2. Slightly too small
  3. Fits well
  4. Slightly too large
  5. Extremely large
Time Frame: 1 day
Measure: Count of Participants; unit: Participants
Arm/Group | Transparent Mask | Non-Transparent Mask
Number analyzed (Participants) | 202 | 202
Participants
  Extremely small | 2 | 4
  Slightly too small | 7 | 29
  Fits well | 172 | 142
  Slightly too large | 21 | 27
  Extremely large | 0 | 0

3. Secondary Outcome: Comfort of the Mask
Description: As recorded on the survey
  1. Not comfortable at all
  2. Slightly comfortable
  3. Very comfortable
  4. Extremely comfortable
Time Frame: 1 day
Measure: Count of Participants; unit: Participants
Arm/Group | Transparent Mask | Non-Transparent Mask
Number analyzed (Participants) | 202 | 202
Participants
  Not comfortable at all | 2 | 31
  Slightly comfortable | 46 | 110
  Very comfortable | 115 | 53
  Extremely comfortable | 39 | 8

4. Secondary Outcome: Ease of Breathing
Description: As recorded on the survey
  1. Not easy at all
  2. Slightly breathable
  3. Very breathable
  4. Extremely breathable
Time Frame: 1 day
Measure: Count of Participants; unit: Participants
Arm/Group | Transparent Mask | Non-Transparent Mask
Number analyzed (Participants) | 202 | 202
Participants
  Not easy at all | 1 | 25
  Slightly breathable | 31 | 85
  Very breathable | 123 | 81
  Extremely breathable | 47 | 11

5. Secondary Outcome: Ease of Speaking/Communicating
Description: As recorded on the survey
  1. Difficult
  2. Somewhat difficult
  3. Somewhat easy
  4. Easy
Time Frame: 1 day
Measure: Count of Participants; unit: Participants
Arm/Group | Transparent Mask | Non-Transparent Mask
Number analyzed (Participants) | 202 | 202
Participants
  Difficult | 0 | 20
  Somewhat difficult | 9 | 64
  Somewhat easy | 36 | 64
  Easy | 157 | 54

ADVERSE EVENTS:
Time Frame: 1 day
Description: Exclusionary criteria were provided and the masks evaluated were not in a clinical environment
Arm/Group | Transparent Mask | Non-Transparent Mask
All-Cause Mortality (participants affected / at risk) | 0/202 | 0/202
Serious Adverse Events (participants affected / at risk) | 0/202 | 0/202
Other Adverse Events (participants affected / at risk) | 0/202 | 0/202

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-01-13): https://cdn.clinicaltrials.gov/large-docs/94/NCT04854694/Prot_000.pdf
  • Statistical Analysis Plan (2023-01-13): https://cdn.clinicaltrials.gov/large-docs/94/NCT04854694/SAP_002.pdf